CLINICAL TRIAL: NCT01963611
Title: A Phase II, Randomized, Multi-center, Parallel-group, Rater-blinded Study to Evaluate the Efficacy, Safety and Tolerability of 0.5 mg, 3 mg, 10 mg and 20 mg Plovamer Acetate Doses Compared to Copaxone in Patients With Relapsing Remitting Multiple Sclerosis
Brief Title: Efficacy, Safety, and Tolerability of Plovamer Acetate (Pathway 1)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated based on sponsor discretion.
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMR200575-001; 2013-002283-25 (EudraCT Number)
Record Dates: First submitted 2013-10-11; First posted 2013-10-16 (Estimated); Results first posted 2016-05-11 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-04

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Multiple Sclerosis; Relapsing Remitting; Plovamer acetate; Copaxone
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Glatiramer Acetate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Plovamer acetate 0.5 milligram (mg) (Experimental): Plovamer acetate was administered at a dose of 0.5 mg as weekly subcutaneous injection for 40 weeks up to a maximum of 14 months.
  Interventions: Drug: Plovamer acetate 0.5 milligram (mg)
- Plovamer acetate 3 mg (Experimental): Plovamer acetate was administered at a dose of 3 mg as weekly subcutaneous injection for 40 weeks up to a maximum of 14 months.
  Interventions: Drug: Plovamer acetate 3 mg
- Plovamer acetate 10 mg (Experimental): Plovamer acetate was administered at a dose of 10 mg as weekly subcutaneous injection for 40 weeks up to a maximum of 14 months.
  Interventions: Drug: Plovamer acetate 10 mg
- Plovamer acetate 20 mg (Experimental): Plovamer acetate was administered as two subcutaneous injection of 10 mg weekly for 40 weeks up to a maximum of 14 months.
  Interventions: Drug: Plovamer acetate 20 mg
- Copaxone 20 mg (Active Comparator): Copaxone was administered at a dose of 20 mg as subcutaneous injection once daily for 40 weeks up to a maximum of 14 months.
  Interventions: Drug: Copaxone 20 mg

INTERVENTIONS:
Drug: Plovamer acetate 0.5 milligram (mg) — Plovamer acetate was administered at a dose of 0.5 mg as weekly subcutaneous injection for 40 weeks up to a maximum of 14 months.
  Arms: Plovamer acetate 0.5 milligram (mg)
Drug: Copaxone 20 mg — Plovamer acetate was administered at a dose of 3 mg as weekly subcutaneous injection for 40 weeks up to a maximum of 14 months.
  Arms: Copaxone 20 mg
Drug: Plovamer acetate 3 mg — Plovamer acetate was administered at a dose of 10 mg as weekly subcutaneous injection for 40 weeks up to a maximum of 14 months.
  Arms: Plovamer acetate 3 mg
Drug: Plovamer acetate 10 mg — Plovamer acetate was administered as two subcutaneous injection of 10 mg weekly for 40 weeks up to a maximum of 14 months.
  Arms: Plovamer acetate 10 mg
Drug: Plovamer acetate 20 mg — Copaxone was administered at a dose of 20 mg as subcutaneous injection once daily for 40 weeks up to a maximum of 14 months.
  Arms: Plovamer acetate 20 mg

SUMMARY:
This is a Phase 2, randomized, rater-blinded, 5-arm, parallel-group trial that will test 4 doses of plovamer acetate against the active comparator Copaxone in subjects with Relapsing Remitting Multiple Sclerosis (RRMS). The trial will be conducted on an outpatient basis for minimum treatment duration of 40 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, between the ages of 18 and 60 years
* Subject is able to learn and self-administer subcutaneous injections (a care-giver may be trained to inject the subject)
* Subjects must have a current diagnosis of Relapsing Remitting Multiple Sclerosis (RRMS) (according to the 2010 McDonald MS diagnostic criteria)
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Any multiple sclerosis categorized as primary progressive, secondary progressive or progressive relapsing
* Allergy to mannitol, plovamer acetate, Copaxone (glatiramer acetate), Gd contrast for MRI
* Any requirement for continuous systemic glucocorticoid administration during the trial period. (Note: Treatment with interferons such as Avonex®, Rebif®, or Betaseron® will be allowed until the baseline visit, as no wash-out period is needed)
* Contraindication to Copaxone use
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 255 (Actual)
Dates: Start 2013-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono, Inc., Billerica MA, a subsidiary of Merck KGaA, Darmstadt, Germany
Locations (117):
- United States (34):
  - Research site, Redding, California
  - Research site, San Diego, California
  - Research site, Fairfield, Connecticut
  - Research site, Dover, Delaware
  - Research site, Miami, Florida
  - Research site, Naples, Florida
  - Research site, Pompano Beach, Florida
  - Research site, Sarasota, Florida
  - Research site, Sunrise, Florida
  - Research site, Columbus, Georgia
  - Research site, Rome, Georgia
  - Research site, Elk Grove Village, Illinois
  - Research site, Indianapolis, Indiana
  - Research site, Baltimore, Maryland
  - Research site, New Bedford, Massachusetts
  - Research site, Worcester, Massachusetts
  - Research site, Detroit, Michigan
  - Research Site, Detroit, Michigan
  - Research site, Golden Valley, Minnesota
  - Research site, St Louis, Missouri
  - Research site, Plainview, New York
  - Research site, Charlotte, North Carolina
  - Research site, Hickory, North Carolina
  - Research site, Matthews, North Carolina
  - Research site, Raleigh, North Carolina
  - Research site, Wilmington, North Carolina
  - Research site, Cincinnati, Ohio
  - Research site, Dayton, Ohio
  - Research site, Willow Grove, Pennsylvania
  - Research site, Nashville, Tennessee
  - Research Site, Round Rock, Texas
  - Research Site, San Antonio, Texas
  - Research site, Roanoke, Virginia
  - Research site, Tacoma, Washington
- Bulgaria (3):
  - Research site, Blagoevgrad
  - Research site, Dupnitsa
  - Research site, Sofia
- Croatia (3):
  - Research site, Osijek
  - Research site, Varaždin
  - Research site, Zagreb
- Czechia (6):
  - Research site, Brno
  - Research site, Havířov
  - Research site, Hradec Králové
  - Research site, Jihlava
  - Research site, Olomouc
  - Research site, Prague
- Finland (3):
  - Research site, Kuopio
  - Research site, Oulu
  - Research site, Turku
- Greece (2):
  - Research site, Athens
  - Research site, Thessaloniki
- Hungary (4):
  - Research site, Budapest
  - Research site, Debrecen
  - Research site, Esztergom
  - Research site, Miskolc
- Italy (8):
  - Research site, Castelfiorentino
  - Research site, Catania
  - Research site, Cefalù
  - Research site, Milan
  - Research site, Modena
  - Research site, Montichiari
  - Research site, Parma
  - Research site, Roma
- Mexico (7):
  - Research site, Cuautitlán Izcalli
  - Research site, León
  - Research site, Mexico City
  - Research site, México
  - Research site, Monterrey
  - Research site, Morelia
  - Research site, Tlalnepantla
- Poland (7):
  - Research site, Gdansk
  - Research site, Katowice
  - Research site, Lodz
  - Research site, Olsztyn
  - Research site, Poznan
  - Research site, Rzeszów
  - Research site, Warsaw
- Russia (10):
  - Research site, Krasnoyarsk
  - Research site, Kursk
  - Research site, Moscow
  - Research site, Nizhny Novgorod
  - Research site, Novosibirsk
  - Research site, Rostov-on-Don
  - Research site, Saint Petersburg
  - Research site, Saransk
  - Research site, Ufa
  - Research site, Yekaterinburg
- Serbia (3):
  - Research site, Belgrade
  - Research site, Kragujevac
  - Research site, Niš
- South Africa (3):
  - Research site, Cape Town
  - Research site, Durban
  - Research site, Pretoria
- Spain (6):
  - Research site, Aranjuez
  - Research site, Córdoba
  - Research site, Madrid
  - Research site, Móstoles
  - Research site, Santander
  - Research site, Zaragoza
- Turkey (Türkiye) (6):
  - Research site, Diyarbakır
  - Research site, Edirne
  - Research site, Istanbul
  - Research site, Kocaeli
  - Research site, Mersin
  - Research site, Samsun
- Ukraine (7):
  - Research site, Dnipropetrovsk
  - Research site, Ivano-Frankivsk
  - Research site, Kyiv
  - Research site, Lutsk
  - Research site, Simferopol
  - Research site, Vinnytsia
  - Research site, Zaporizhzhia
- United Kingdom (5):
  - Research site, Exeter
  - Research site, Hull
  - Research site, Sheffield
  - Research site, Southampton
  - Research site, Stoke-on-Trent

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Plovamer Acetate 0.5 Milligram (mg) | Plovamer Acetate 3 mg | Plovamer Acetate 10 mg | Plovamer Acetate 20 mg | Copaxone 20 mg
Started | 51 | 49 | 52 | 52 | 51
Safety Analysis Set | 51 | 49 | 52 | 52 | 50
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 51 | 49 | 52 | 52 | 51
Not completed — Adverse Event | 1 | 1 | 3 | 4 | 3
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 1 | 1 | 3
Not completed — Other | 47 | 46 | 48 | 45 | 45

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAF) includes all randomized subjects who had received at least 1 dose of investigational medicinal product (IMP).
Groups:
- Total: Total of all reporting groups
Arm/Group | Plovamer Acetate 0.5 Milligram (mg) | Plovamer Acetate 3 mg | Plovamer Acetate 10 mg | Plovamer Acetate 20 mg | Copaxone 20 mg | Total
Number analyzed (Participants) | 51 | 49 | 52 | 52 | 50 | 254
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (10.73) | 40.7 (9.54) | 41.1 (10.83) | 40.4 (9.53) | 41.8 (11.61) | 40.6 (10.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 37 | 39 | 37 | 26 | 177
  Male | 13 | 12 | 13 | 15 | 24 | 77

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Time Constant 1 (T1) Gadolinium (Gd)-Enhancing Lesions Per Subject and Scan
Description: Time Constant 1 (T1) Gadolinium (Gd)-Enhancing Lesions per Subject and Scan was calculated using 5 serial magnetic resonance imaging (MRI) scans.
Time Frame: Baseline , Week 12, 24, 28, 32, 36, 40
Population: Intent to Treat (ITT) analysis set included all randomized subjects with at least 1 post-baseline efficacy (MRI) assessment. Here 'n' signifies those participants who were evaluated for this measure at the specified time point for each arm group respectively.
Measure: Mean (Standard Deviation); unit: lesions per subjects per scan
Arm/Group | Plovamer Acetate 0.5 Milligram (mg) | Plovamer Acetate 3 mg | Plovamer Acetate 10 mg | Plovamer Acetate 20 mg | Copaxone 20 mg
Number analyzed (Participants) | 45 | 45 | 43 | 41 | 44
lesions per subjects per scan
  Baseline (n=44,45,42,41,44) | 1.5 (2.93) | 1.6 (4.12) | 1.0 (2.43) | 2.3 (5.65) | 2.5 (5.12)
  Week 12: (n=44,45,43,41,44) | 1.7 (3.28) | 1.3 (3.55) | 1.2 (2.40) | 1.5 (3.70) | 1.7 (4.51)
  Week 24: (n=17,17,21,18,19) | 1.5 (2.53) | 0.9 (2.33) | 1.5 (4.14) | 1.1 (1.92) | 0.6 (1.46)
  Week 28: (n=10,11,13,12,13) | 1.7 (2.75) | 0.4 (0.92) | 0.5 (1.20) | 2.0 (4.00) | 0.9 (1.89)
  Week 32: (n=5,6,9,10,9) | 1.0 (1.41) | 0.2 (0.41) | 0.8 (1.72) | 1.8 (3.33) | 1.2 (3.67)
  Week 36: (n=1,0,2,3,3) | 0.0 (NA) — Standard deviation was not reported as number of subject analyzed was 1. | NA (NA) — Data was not reported as there was no subject. | 1.0 (1.41) | 1.3 (2.31) | 7.3 (12.70)
  Week 40: (n=1,0,1,1,1) | 0.0 (NA) — Standard deviation was not reported as number of subject analyzed was 1. | NA (NA) — Data was not reported as there was no subject. | 0.0 (NA) — Standard deviation was not reported as number of subject analyzed was 1. | 0.0 (NA) — Standard deviation was not reported as number of subject analyzed was 1. | 16.0 (NA) — Standard deviation was not reported as number of subject analyzed was 1.

2. Secondary Outcome: Mean Annualized Relapse Rate (ARR)
Description: Relapse was defined as new, worsening or recurrent neurological symptoms attributed to multiple sclerosis that last for at least 24 hours without fever or infection, or adverse reaction to prescribed medication, preceded by a stable or improving neurological status of at least 30 days. These new or worsening symptoms should be noted by the patient and must be accompanied by at least one of the following: An increase of greater than or equal to (>=) 1 grade in >=2 functional scales of the Expanded Disability Status Scale (EDSS) or an increase of >=2 grades in 1 functional scale of the EDSS or an increase of >= 0.5 or an increase of >=1.0 in EDSS if the previous EDSS was 0. Annualized Relapse Rate was calculated as = 365.25 x (Number of relapses during Treatment Period) per (Number of days on treatment during Treatment Period).
Time Frame: Baseline up to Week 40
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percent relapse
Arm/Group | Plovamer Acetate 0.5 Milligram (mg) | Plovamer Acetate 3 mg | Plovamer Acetate 10 mg | Plovamer Acetate 20 mg | Copaxone 20 mg
Number analyzed (Participants) | 51 | 49 | 52 | 52 | 50
percent relapse | 0.3 (0.88) | 0.2 (0.62) | 0.2 (0.76) | 0.2 (0.88) | 0.2 (0.92)

3. Secondary Outcome: Percentage of Subjects Remaining Relapse-Free
Description: Relapse was defined as new, worsening or recurrent neurological symptoms attributed to multiple sclerosis that last for at least 24 hours without fever or infection, or adverse reaction to prescribed medication, preceded by a stable or improving neurological status of at least 30 days. These new or worsening symptoms should be noted by the patient and must be accompanied by at least one of the following: An increase of greater than or equal to (>=) 1 grade in >=2 functional scales of the Expanded Disability Status Scale (EDSS) or an increase of >=2 grades in 1 functional scale of the EDSS or an increase of >= 0.5 or an increase of >=1.0 in EDSS if the previous EDSS was 0.
Time Frame: Baseline up to Week 40
Population: as for baseline characteristics
Measure: Number; unit: percent subjects
Arm/Group | Plovamer Acetate 0.5 Milligram (mg) | Plovamer Acetate 3 mg | Plovamer Acetate 10 mg | Plovamer Acetate 20 mg | Copaxone 20 mg
Number analyzed (Participants) | 51 | 49 | 52 | 52 | 50
percent subjects | 86.3 | 89.8 | 94.2 | 94.2 | 90.0

4. Secondary Outcome: Mean Number of New T1 Gadolinium (Gd)-Enhancing Lesions Per Subject and Scan
Description: T1 Gd-enhancing lesions per subject and scan was measured using 5 serial MRI scans.
Time Frame: Weeks 12, 24, 28, 32, 36, 40
Population: ITT analysis set included all randomized subjects with at least 1 post-baseline efficacy (MRI) assessment. Here "n" signifies those participants who were evaluated for this measure at the specified time point for each arm group respectively.
Measure: Mean (Standard Deviation); unit: lesions/subject/scan
Arm/Group | Plovamer Acetate 0.5 Milligram (mg) | Plovamer Acetate 3 mg | Plovamer Acetate 10 mg | Plovamer Acetate 20 mg | Copaxone 20 mg
Number analyzed (Participants) | 45 | 45 | 43 | 41 | 44
lesions/subject/scan
  Week 12: (n=44,45,43,41,44) | 1.7 (3.26) | 1.2 (3.54) | 1.2 (2.26) | 1.3 (2.99) | 1.6 (4.31)
  Week 24: (n=17,17,21,18,19) | 1.5 (2.53) | 0.9 (2.33) | 1.4 (3.56) | 1.0 (1.94) | 0.5 (1.26)
  Week 28: (n=10,11,13,12,13) | 1.2 (2.15) | 0.1 (0.30) | 0.5 (1.13) | 1.8 (3.83) | 0.5 (1.33)
  Week 32: (n=5,6,9,10,9) | 0.8 (1.10) | 0.2 (0.41) | 0.4 (1.33) | 1.5 (2.95) | 0.6 (1.67)
  Week 36: (n=1,0,2,3,3) | 0.0 (NA) — Standard deviation was not reported as number of subject analyzed was 1. | NA (NA) — Data was not reported as there was no subject. | 0.5 (0.71) | 1.0 (1.73) | 5.7 (9.81)
  Week 40: (n=1,0,1,1,1) | 0.0 (NA) — Standard deviation was not reported as number of subject analyzed was 1. | NA (NA) — Data was not reported as there was no subject. | 0.0 (NA) — Standard deviation was not reported as number of subject analyzed was 1. | 0.0 (NA) — Standard deviation was not reported as number of subject analyzed was 1. | 16.0 (NA) — Standard deviation was not reported as number of subject analyzed was 1.

5. Secondary Outcome: Mean Number of New or Enlarging Time Constant 2 (T2) Lesions Per Subject and Scan
Description: New or enlarging Time Constant 2 (T2) lesions per subject and scan was calculated using 5 serial MRI scans.
Time Frame: Weeks 12, 24, 28, 32, 36,40
Population: ITT analysis set included all randomized subjects with at least 1 post-baseline efficacy (MRI) assessment. Here 'n' signifies those participants who were evaluated for this measure at the specified time point for each arm group respectively.
Measure: Mean (Standard Deviation); unit: lesions/subject/scan
Arm/Group | Plovamer Acetate 0.5 Milligram (mg) | Plovamer Acetate 3 mg | Plovamer Acetate 10 mg | Plovamer Acetate 20 mg | Copaxone 20 mg
Number analyzed (Participants) | 45 | 45 | 43 | 41 | 44
lesions/subject/scan
  Week 12: (n=44,45,43,41,44) | 4.5 (7.41) | 2.6 (4.99) | 2.7 (4.50) | 4.1 (7.45) | 4.0 (8.59)
  Week 24: (n=17,17,21,18,19) | 3.1 (5.61) | 1.8 (3.35) | 2.3 (4.91) | 3.4 (6.03) | 1.7 (3.45)
  Week 28: (n=10,11,13,12,13) | 1.3 (2.45) | 0.2 (0.40) | 0.8 (1.69) | 2.5 (5.05) | 0.8 (2.15)
  Week 32: (n=5,6,9,10,9) | 1.4 (2.19) | 0.2 (0.41) | 0.3 (0.71) | 2.4 (4.12) | 0.9 (2.32)
  Week 36: (n=1,0,2,3,3) | 0.0 (NA) — Standard deviation was not reported as number of subject analyzed was 1. | NA (NA) — Data was not reported as there was no subject. | 0.5 (0.71) | 1.7 (2.89) | 4.3 (7.51)
  Week 40: (n=1,0,1,1,1) | 0.0 (NA) — Standard deviation was not reported as number of subject analyzed was 1. | NA (NA) — Data was not reported as there was no subject. | 0.0 (NA) — Standard deviation was not reported as number of subject analyzed was 1. | 0.0 (NA) — Standard deviation was not reported as number of subject analyzed was 1. | 13.0 (NA) — Standard deviation was not reported as number of subject analyzed was 1.

6. Secondary Outcome: Mean Number of New, Unenhancing T1 Lesions (Black Holes) Per Subject and Scan
Description: New, unenhancing T1 lesions (Black Holes) per subject and scan was calculated using 5 Serial MRIs.
Time Frame: Weeks 12, 24, 28, 32, 36, 40
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: lesions/subject/scan
Arm/Group | Plovamer Acetate 0.5 Milligram (mg) | Plovamer Acetate 3 mg | Plovamer Acetate 10 mg | Plovamer Acetate 20 mg | Copaxone 20 mg
Number analyzed (Participants) | 45 | 45 | 43 | 41 | 44
lesions/subject/scan
  Week 12: (n=44,45,43,41,44) | 2.8 (6.48) | 1.8 (3.97) | 1.4 (2.21) | 2.6 (5.24) | 2.6 (5.13)
  Week 24: (n=17,17,21,18,19) | 2.0 (4.80) | 0.8 (1.55) | 0.8 (1.83) | 1.3 (2.89) | 0.8 (1.75)
  Week 28: (n=10,11,13,12,13) | 0.6 (1.26) | 0.2 (0.60) | 0.6 (1.56) | 0.5 (1.00) | 0.4 (1.39)
  Week 32: (n=5,6,9,10,9) | 2.0 (3.39) | 0.2 (0.41) | 0.8 (1.30) | 0.7 (1.25) | 0.3 (0.71)
  Week 36: (n=1,0,2,3,3) | 0.0 (NA) — Standard deviation was not reported as number of subject analyzed was 1. | NA (NA) — Data was not reported as there was no subject. | 0.0 (0.00) | 0.7 (1.15) | 1.7 (2.89)
  Week 40: (n=1,0,1,1,1) | 0.0 (NA) — Standard deviation was not reported as number of subject analyzed was 1. | NA (NA) — Data was not reported as there was no subject. | 0.0 (NA) — Standard deviation was not reported as number of subject analyzed was 1. | 0.0 (NA) — Standard deviation was not reported as number of subject analyzed was 1. | 11.0 (NA) — Standard deviation was not reported as number of subject analyzed was 1.

7. Secondary Outcome: Mean Change From Baseline in Volume of T1 Gadolinium (Gd)-Enhancing Lesions Per Subject and Scan
Description: Change from baseline in volume of T1 Gd-enhancing lesions per subject was calculated using 5 Serial MRI Scans.
Time Frame: Baseline, Weeks 12, 24, 28, 32, 36, 40
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: cubic millimeter (mm^3)
Arm/Group | Plovamer Acetate 0.5 Milligram (mg) | Plovamer Acetate 3 mg | Plovamer Acetate 10 mg | Plovamer Acetate 20 mg | Copaxone 20 mg
Number analyzed (Participants) | 45 | 45 | 43 | 41 | 44
cubic millimeter (mm^3)
  Baseline: (n=44,45,42,41,44) | 0.182 (0.4212) | 0.209 (0.6325) | 0.138 (0.3577) | 0.508 (1.1981) | 0.264 (0.5707)
  Change at Week 12: (n=44,45,42,41,44) | 0.037 (0.3982) | -0.007 (0.6019) | 0.189 (0.8406) | -0.190 (1.0389) | 0.023 (0.5794)
  Change at Week 24: (n=16,17,20,18,19) | 0.053 (0.1705) | 0.352 (1.4308) | 0.060 (0.4858) | -0.591 (1.4910) | -0.250 (0.5393)
  Change at Week 28: (n=9,11,12,12,13) | 0.224 (0.2948) | 0.067 (0.4640) | 0.057 (0.5728) | -0.796 (1.7779) | -0.257 (0.6980)
  Change at Week 32: (n=4,6,8,10,9) | -0.085 (0.2765) | -0.102 (0.2691) | -0.135 (0.6305) | -0.988 (1.9800) | 0.031 (0.8312)
  Change at Week 36: (n=0,0,1,3,3) | NA (NA) — Data was not reported as there was no subject. | NA (NA) — Data was not reported as there was no subject. | 0.321 (NA) — Standard deviation was not reported as number of subject analyzed was 1. | -1.881 (3.4679) | 0.834 (2.1816)
  Change at Week 40: (n=0,0,0,1,1) | NA (NA) — Data was not reported as there was no subject. | NA (NA) — Data was not reported as there was no subject. | NA (NA) — Data was not reported as there was no subject. | 0.000 (NA) — Standard deviation was not reported as number of subject analyzed was 1. | 2.180 (NA) — Standard deviation was not reported as number of subject analyzed was 1.

8. Secondary Outcome: Mean Change From Baseline in Volume of T2 Gadolinium (Gd)-Enhancing Lesions Per Subject and Scan
Description: Change from baseline per subjects in volume of T2 Gd-enhancing lesions was calculated using 5 series MRI scan.
Time Frame: Baseline, Weeks 12, 24, 28, 32, 36, 40
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: cubic millimeter (mm^3)
Arm/Group | Plovamer Acetate 0.5 Milligram (mg) | Plovamer Acetate 3 mg | Plovamer Acetate 10 mg | Plovamer Acetate 20 mg | Copaxone 20 mg
Number analyzed (Participants) | 45 | 45 | 43 | 41 | 44
cubic millimeter (mm^3)
  Baseline (n=44,45,42,41,44) | 12.240 (14.6956) | 13.482 (19.0522) | 11.364 (16.0282) | 9.518 (13.2248) | 11.616 (15.4960)
  Change at Week 12: (n=44,45,42,41,44) | 0.443 (2.2414) | 0.397 (1.0399) | 0.686 (2.4894) | -0.200 (4.5312) | 0.060 (1.3886)
  Change at Week 24: (n=16,17,20,18,19) | -0.179 (2.2741) | 0.871 (2.7803) | 0.113 (1.2011) | -1.734 (6.8085) | -0.907 (2.5627)
  Change at Week 28: (n=9,11,12,12,13) | 0.016 (3.2248) | 0.858 (3.0417) | 0.306 (1.1945) | -2.610 (8.3108) | -1.379 (3.4251)
  Change at Week 32: (n=4,6,8,10,9) | 0.874 (2.4859) | 0.163 (1.2524) | -0.106 (1.3423) | -3.246 (9.3533) | -1.867 (3.6432)
  Change at Week 36: (n=0,0,1,3,3) | NA (NA) — Data was not reported as there was no subject. | NA (NA) — Data was not reported as there was no subject. | 1.236 (NA) — Standard deviation was not reported as number of subject analyzed was 1. | -10.324 (17.2227) | -4.433 (4.6895)
  Change at Week 40: (n=0,0,0,1,1) | NA (NA) — Data was not reported as there was no subject. | NA (NA) — Data was not reported as there was no subject. | NA (NA) — Data was not reported as there was no subject. | -29.965 (NA) — Standard deviation was not reported as number of subject analyzed was 1. | -10.661 (NA) — Standard deviation was not reported as number of subject analyzed was 1.

9. Secondary Outcome: Time to First Relapse
Description: as for outcome 3
Time Frame: Baseline up to Week 40
Population: The Outcome Measure was not derived due to early termination of the study.
Arm/Group | Plovamer Acetate 0.5 Milligram (mg) | Plovamer Acetate 3 mg | Plovamer Acetate 10 mg | Plovamer Acetate 20 mg | Copaxone 20 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Mean Change From Baseline in Brain Volume Per Subject
Description: Change from baseline in brain volume per subject was calculated using 5 series MRI scan.
Time Frame: Baseline, Weeks 24, 28, 32, 36, 40
Population: The Outcome Measure was not derived due to early termination of the study.
Arm/Group | Plovamer Acetate 0.5 Milligram (mg) | Plovamer Acetate 3 mg | Plovamer Acetate 10 mg | Plovamer Acetate 20 mg | Copaxone 20 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to end of treatment (week 40)
Groups:
- Plovamer Acetate 0.5 Milligram (mg): Plovamer acetate was administered at a dose of 0.5 mg as weekly subcutaneous injection for a minimum of 40 weeks.
- Plovamer Acetate 3 mg: Plovamer acetate was administered at a dose of 3 mg as weekly subcutaneous injection for a minimum of 40 weeks.
- Plovamer Acetate 10 mg: Plovamer acetate was administered at a dose of 10 mg as weekly subcutaneous injection for a minimum of 40 weeks.
- Plovamer Acetate 20 mg: Plovamer acetate was administered at a dose of 20 mg as weekly subcutaneous injection for a minimum of 40 weeks.
- Copaxone 20 mg: Copaxone was administered at a dose of 20 mg as subcutaneous injection once daily for a minimum of 40 weeks.
Arm/Group | Plovamer Acetate 0.5 Milligram (mg) | Plovamer Acetate 3 mg | Plovamer Acetate 10 mg | Plovamer Acetate 20 mg | Copaxone 20 mg
Serious Adverse Events (participants affected / at risk) | 2/51 | 0/49 | 2/52 | 3/52 | 0/50
Other Adverse Events (participants affected / at risk) | 28/51 | 34/49 | 38/52 | 41/52 | 42/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Plovamer Acetate 0.5 Milligram (mg) (N=51) | Plovamer Acetate 3 mg (N=49) | Plovamer Acetate 10 mg (N=52) | Plovamer Acetate 20 mg (N=52) | Copaxone 20 mg (N=50)
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Plovamer Acetate 0.5 Milligram (mg) (N=51) | Plovamer Acetate 3 mg (N=49) | Plovamer Acetate 10 mg (N=52) | Plovamer Acetate 20 mg (N=52) | Copaxone 20 mg (N=50)
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 6 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 3 | 4
Urinary tract infection (Infections and infestations) | 2 | 0 | 1 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 2 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 2 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Erythema migrans (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Chronic tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Tracheitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urethritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 1 | 2 | 0 | 0
Depressive symptom (Psychiatric disorders) | 0 | 2 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0
Adjustment disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Affective disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1
Emotional disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Mood altered (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Nightmare (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 4 | 0 | 1 | 4 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 2 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Essential tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Muscle spasticity (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Radicular pain (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Perineurial cyst (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Eyelid skin dryness (Eye disorders) | 0 | 0 | 0 | 1 | 0
Iritis (Eye disorders) | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 2 | 2 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Melanosis coli (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal rigidity (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Myokymia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Epididymal cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Injection site pain (General disorders) | 8 | 20 | 26 | 26 | 28
Injection site erythema (General disorders) | 10 | 16 | 14 | 19 | 18
Injection site pruritus (General disorders) | 3 | 6 | 10 | 4 | 15
Injection site induration (General disorders) | 1 | 2 | 5 | 6 | 4
Injection site oedema (General disorders) | 1 | 1 | 2 | 2 | 2
Injection site bruising (General disorders) | 3 | 1 | 0 | 1 | 3
Influenza like illness (General disorders) | 1 | 1 | 1 | 0 | 1
Injection site haematoma (General disorders) | 1 | 0 | 0 | 2 | 4
Injection site laceration (General disorders) | 0 | 1 | 1 | 1 | 0
Injection site nodule (General disorders) | 0 | 1 | 2 | 0 | 0
Injection site rash (General disorders) | 1 | 0 | 1 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 2 | 0
Asthenia (General disorders) | 0 | 1 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 1 | 0
Chills (General disorders) | 0 | 1 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 0 | 1
Injection site haemorrhage (General disorders) | 0 | 0 | 0 | 2 | 0
Injection site paraesthesia (General disorders) | 1 | 0 | 1 | 0 | 0
Injection site swelling (General disorders) | 0 | 0 | 1 | 1 | 1
Oedema peripheral (General disorders) | 0 | 1 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 1 | 0 | 0
Injection site cyst (General disorders) | 0 | 0 | 0 | 1 | 0
Injection site mass (General disorders) | 0 | 0 | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 0 | 1 | 0 | 0
Cyst (General disorders) | 0 | 0 | 0 | 0 | 1
Hyperthermia (General disorders) | 0 | 0 | 0 | 0 | 1
Injection site discolouration (General disorders) | 0 | 0 | 0 | 0 | 1
Injection site granuloma (General disorders) | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Electrocardiogram PR shortened (Investigations) | 0 | 1 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Based on Sponsor decision to discontinue the clinical development program of plovamer acetate therapy for multiple sclerosis the trial was prematurely terminated

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other